CLINICAL TRIAL: NCT04385225
Title: Effect of Hearing Loss and Vestibular Decline on Cognitive Function in Older Subjects: Correlation With Cortical Auditory Evoked Potentials and MRI Brain Volume Changes
Brief Title: Effect of Hearing Loss and Vestibular Decline on Cognitive Function in Older Subjects
Acronym: GECkO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, Prof. dr. Vincent Van Rompaey, principal investigator, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B300201938949
Record Dates: First submitted 2020-02-03; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Hearing Loss, Sensorineural; Bilateral Vestibulopathy; Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Hearing Loss, Sensorineural; Bilateral Vestibulopathy; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy controls (Other): Age-matched controls with normal hearing or mild sensorineural hearing loss: 40 decibel or less in better hearing ear, and normal vestibular function
  Interventions: Other: Longitudinal follow-up
- Moderate Sensorineural hearing loss (Other): Moderate Sensorineural hearing loss: 41-60 decibel in the better hearing ear
  Interventions: Other: Longitudinal follow-up
- Severe Sensorineural hearing loss (Other): Severe Sensorineural hearing loss: 61-80 decibel in the better hearing ear
  Interventions: Other: Longitudinal follow-up
- Bilateral Vestibulopathy (Other): Bilateral vestibulopathy: half with normal hearing, half with severe to profound sensorineural hearing loss
  Interventions: Other: Longitudinal follow-up
- Mild Cognitive Impairment (Other): Mild Cognitive Impairment
  Interventions: Other: Longitudinal follow-up
- Alzheimer's Disease (Other): Alzheimer's Disease
  Interventions: Other: Longitudinal follow-up

INTERVENTIONS:
Other: Longitudinal follow-up — Longitudinal hearing, vestibular and cognitive follow-up

SUMMARY:
The world population has been growing and aging dramatically, with a rising prevalence of dementia. Worldwide, around 50 million people have dementia, with 10 million new cases added every year. Despite the epidemic scale of dementia, until now no cure or disease-modifying therapy has been identified. Therefore, the World Health Organization (WHO) has recognized dementia as a public health priority. Several large studies have demonstrated that hearing impairment is associated with a greater risk of cognitive impairment. Hearing rehabilitation could potentially provide a disease-modifying therapy to delay cognitive decline. Although auditory behavioral research has not yet revealed a reliable indicator of early cognitive impairment, cortical-evoked auditory potentials (CAEP) have shown promising evidence as a non-invasive way to identify early-stage cognitive impairment.

The peripheral vestibular apparatus is located in the inner ear and codes rotation and translation of the head to preserve a stable view. Increasing evidence suggests that bilateral vestibular function loss, also known as bilateral vestibulopathy (BVP), leads to hippocampal atrophy and reduced spatial cognitive skills, as well as structural and functional alterations in parieto-insular and parieto-temporal regions. Many studies have demonstrated that vestibular function declines with age. Vestibular dysfunction can be linked to reduced topographical orientation and memory and has been suggested as a risk factor to AD, due to increased risk of falling and deficits in activities of daily life (ADL).

Our first aim is to study the effect of SNHL and vestibular decline on CAEP, spatial and non-spatial cognitive functioning and trajectories in cognitively healthy older subjects, as well as patients with mild cognitive impairment (MCI) and AD. Our second aim is to study if MRI brain volume changes can be observed in the hippocampus, entorhinal cortex, and auditory and vestibular key regions in these populations and correlate with CAEP and cognitive functioning.

The expected outcome is important to society because it will provide data from a cognitive assessment protocol adapted for a potentially hearing-impaired population, objective outcome measures (incl. CAEP and MRI brain volume changes) to identify older subjects with SNHL and BVP at risk for cognitive decline, and will support screening and interventional studies to assess the impact of rehabilitation on slowing down cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination > 12
* Dutch-speaking

Exclusion Criteria:

* Uncorrectable visual impairment
* Hearing implants
* Hearing aids

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals total score | Longitudinal follow-up for 24 months
  Cognitive test adapted for hearing impaired subjects, minimum score is 200, maximum score is 800, higher scores indicate better cognitive performance

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bosmans J, Jorissen C, Cras P, Van Ombergen A, Engelborghs S, Gilles A, Princen E, Moyaert J, Mertens G, Van Rompaey V. Impact of hearing loss and vestibular decline on cognition in Alzheimer's disease: a prospective longitudinal study protocol (Gehoor, Evenwicht en Cognitie, GECkO). BMJ Open. 2020 Sep 17;10(9):e039601. doi: 10.1136/bmjopen-2020-039601. PMID 32948575